CLINICAL TRIAL: NCT01493414
Title: An Open-label, Multicenter, Expanded Access Study of INC424 for Patients With Primary Myelofibrosis (PMF) or Post Polycythemia Myelofibrosis (PPV MF) or Post-essential Thrombocythemia Myelofibrosis (PET-MF).
Brief Title: INC424 for Patients With Primary Myelofibrosis, Post Polycythemia Myelofibrosis or Post-essential Thrombocythemia Myelofibrosis.
Acronym: JUMP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC424A2401; 2010-024473-39 (EudraCT Number)
Record Dates: First submitted 2011-12-13; First posted 2011-12-16 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2018-10

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Primary myelofibrosis; PMF; Post polycythemia myelofibrosis; PPV MF; Post-essential thrombocythemia myelofibrosis; PET-MF; INC424; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INC424 (Experimental): 5 - 25 mg twice a day (BID)
  Interventions: Drug: INC424

INTERVENTIONS:
Drug: INC424 — All patients enrolled into the study will receive INC424 (ruxolitinib). Starting dose is based on baseline platelet counts, with doses ranging from 5 to 20 mg twice a day. No INC424 dose will exceed 25 mg BID orally.
  Other Names: Ruxolitinib

SUMMARY:
The primary objective of this study was to collect additional safety of INC424 in patients with Primary Myelofibrosis, Post Polycythemia Myelofibrosis or Post-essential Thrombocythemia Myelofibrosis, who either received prior treatment with commercially available agents or who have never received treatment.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patients must not be eligible for another ongoing INC424 clinical trial.
2. Patients must be diagnosed with PMF, PPV MF or PET-MF, according to the 2008 revised International Standard Criteria, irrespective of JAK2 mutation status..
3. Patients with PMF requiring therapy must be classified as high risk (3 prognostic factors) OR intermediate risk level 2 (2 prognostic factors, no more), OR intermediate risk level 1 (1 prognostic factor, no more) with an enlarged spleen (assessment to occur at the Screening Visit).

   The prognostic factors, defined by the International Working Group are:
   * Age > 65 years;
   * Presence of constitutional symptoms (weight loss, fever, night sweats);
   * Marked anemia (Hgb < 10g/dL)*;
   * Leukocytosis (history of white blood cell (WBC) > 25 x109/L);
   * Circulating blasts > 1%. * A hemoglobin value < 10 g/dL must be demonstrated during the Screening Visit for patients who are not transfusion dependent. Patients receiving regular transfusions of packed red blood cells will be considered to have hemoglobin < 10 g/dL for the purpose of evaluation of risk factors.
4. Patients with Intermediate-1 disease and splenomegaly must have a palpable spleen measuring 5 cm or greater from the costal margin to the point of greatest splenic protrusion.
5. Patients must have a peripheral blood blast count of < 10%.
6. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
7. Fedratinib pretreated patients with documented complete physical examination including full neurologic examination and cardiology assessment, thiamine level testing, and MRI of the brain if indicated based on signs or symptoms. Patients pretreated with fedratinib should have completed or be receiving thiamine supplementation according to the investigator's instructions.

Main Exclusion Criteria:

1. Patients eligible for hematopoietic stem cell transplantation (suitable candidate and a suitable donor is available).
2. Patients with history of malignancy in past 3 years except for treated, early-stage squamous or basal cell carcinoma in situ.
3. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral INC424 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection).
4. Patients with cardiac disease which in the Investigator's opinion may jeopardize the safety of the patient or the compliance with the protocol.
5. Patients with currently uncontrolled or unstable angina, rapid or paroxysmal atrial fibrillation or recent (approximately 6 months) myocardial infarction or acute coronary syndrome.
6. Patients with clinically significant bacterial, fungal, parasitic or viral infection which require therapy. Patients with acute bacterial infections requiring antibiotic use should delay screening/enrollment until the course of antibiotic therapy has been completed.
7. Patients with known active hepatitis A, B, C or who are HIV-positive.
8. Patients with inadequate bone marrow reserve at the Baseline visit as demonstrated by:

   * Absolute neutrophil count (ANC) ≤ 1000/µL.
   * Platelet count < 50,000/µL without the assistance of growth factors, thrombopoietic factors or platelet transfusions.
9. Patients with any history of platelet counts < 50,000/µL or ANC < 500/µL except during treatment for a myeloproliferative disorder or treatment with cytotoxic therapy for any other reason.
10. In the case of ruxolitinib pretreated patients, ruxolitinib primary resistant patients defined as:

    • No spleen reduction within the first 12 weeks after front line therapy with ruxolitinib.

    AND

    • No reduction in symptoms within the first 12 weeks after first-line treatment with ruxolitinib.
11. In the case of ruxolitinib pretreated patients, patients discontinuing ruxolitinib due to a Grade 4 Adverse event (AE) related or suspected to be related to ruxolitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2233 (Actual)
Dates: Start 2011-08-16; Primary Completion 2017-01-26 (Actual); Study Completion 2017-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (232):
- Novartis Investigative Site, Algiers, Algeria
- Argentina (5):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Paraná, Entre Ríos Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
- Austria (5):
  - Novartis Investigative Site, Innsbruck, Tyrol
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (14):
  - Novartis Investigative Site, Arlon, Luxembourg
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Kortrijk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Roeselare
  - Novartis Investigative Site, Wilrijk
  - Novartis Investigative Site, Yvoir
- Brazil (8):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (12):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Windsor, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Colombia (2):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Medellín
- Czechia (4):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Hradec Králové, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Olomouc
- Germany (47):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Bottrop
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt (Oder)
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Friedrichshafen
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hamm
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Ingolstadt
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Leer
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Minden
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Pátrai
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szombathely
- Novartis Investigative Site, Cork, Cork, Ireland
- Israel (6):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (46):
  - Novartis Investigative Site, Alessandria, AL
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pesaro, PU
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Rionero in Vulture, PZ
  - Novartis Investigative Site, Ravenna, RA
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Pagani, SA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Taranto, TA
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Treviso, TV
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Varese, VA
  - Novartis Investigative Site, Venezia, VE
  - Novartis Investigative Site, Vicenza, VI
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Ronciglione, VT
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Perugia
- Mexico (5):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Hermosillo, Sonora
  - Novartis Investigative Site, Puebla City
- Novartis Investigative Site, Marrakesh, Morocco
- Poland (6):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Opole
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
- Portugal (5):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Faro
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Real
- Russia (6):
  - Novartis Investigative Site, Irkutsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
- Saudi Arabia (2):
  - Novartis Investigative Site, Jeddah
  - Novartis Investigative Site, Riyadh
- Novartis Investigative Site, Bratislava, Slovakia
- South Africa (4):
  - Novartis Investigative Site, Soweto, Gauteng
  - Novartis Investigative Site, Cape Town, Western Province
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Pretoria
- Spain (38):
  - Novartis Investigative Site, Ferrol, A Coruna
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Jaén, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Burgos, Castille and León
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Toledo, Castille-La Mancha
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Girona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Logroño, La Rioja
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, Alcalá de Henares, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, San Sebastián de los Reyes, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Zaragoza
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Tunisia (3):
  - Novartis Investigative Site, Sfax, Tunisie
  - Novartis Investigative Site, Sousse
  - Novartis Investigative Site, Tunis

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gupta V, Griesshammer M, Martino B, Foltz L, Tavares R, Al-Ali HK, Giraldo P, Guglielmelli P, Lomaia E, Bouard C, Paley C, Tiwari R, Zor E, Raanani P. Analysis of predictors of response to ruxolitinib in patients with myelofibrosis in the phase 3b expanded-access JUMP study. Leuk Lymphoma. 2021 Apr;62(4):918-926. doi: 10.1080/10428194.2020.1845334. Epub 2020 Nov 19. PMID 33210570
- [Derived] Al-Ali HK, Griesshammer M, Foltz L, Palumbo GA, Martino B, Palandri F, Liberati AM, le Coutre P, Garcia-Hernandez C, Zaritskey A, Tavares R, Gupta V, Raanani P, Giraldo P, Hanel M, Damiani D, Sacha T, Bouard C, Paley C, Tiwari R, Mannelli F, Vannucchi AM. Primary analysis of JUMP, a phase 3b, expanded-access study evaluating the safety and efficacy of ruxolitinib in patients with myelofibrosis, including those with low platelet counts. Br J Haematol. 2020 Jun;189(5):888-903. doi: 10.1111/bjh.16462. Epub 2020 Feb 4. PMID 32017044
- [Derived] Tavares R, Souza CA, Paley C, Bouard C, Tiwari R, Pasquini R. A subgroup analysis of JUMP, a phase IIIb, expanded-access study evaluating the safety and efficacy of ruxolitinib in patients with myelofibrosis in a Brazilian cohort. Hematol Transfus Cell Ther. 2020 Jan-Mar;42(1):46-53. doi: 10.1016/j.htct.2019.01.009. Epub 2019 Apr 25. PMID 31235325
- [Derived] Al-Ali HK, Griesshammer M, le Coutre P, Waller CF, Liberati AM, Schafhausen P, Tavares R, Giraldo P, Foltz L, Raanani P, Gupta V, Tannir B, Ronco JP, Ghosh J, Martino B, Vannucchi AM. Safety and efficacy of ruxolitinib in an open-label, multicenter, single-arm phase 3b expanded-access study in patients with myelofibrosis: a snapshot of 1144 patients in the JUMP trial. Haematologica. 2016 Sep;101(9):1065-73. doi: 10.3324/haematol.2016.143677. Epub 2016 May 31. PMID 27247324

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an expanded access study intended to provide an access path to ruxolitinib for patients with Myelofibrosis (MF) and to allow for collection of additional safety and efficacy data for ruxolitinib.
Period: Overall Study
Arm/Group | INC424
Started | 2233
Completed | 1283
Not Completed | 950
Not completed — Adverse Event | 405
Not completed — Disease progression | 204
Not completed — Death | 101
Not completed — Physician Decision | 93
Not completed — Withdrawal by Subject | 79
Not completed — Protocol deviation | 27
Not completed — Administrative problems | 25
Not completed — Lost to Follow-up | 16

BASELINE CHARACTERISTICS:
Arm/Group | INC424
Number analyzed (Participants) | 2233
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1016
  Male | 1217
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 20
  White | 2087
  More than one race | 96
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 509
  Chinese | 1
  Indian (Indian subcontinent) | 1
  Japanese | 0
  Mixed Ethnicity | 15
  Others | 1707
ECOG score [Count of Participants; unit: Participants] — ECOG Performance Score has 5 grades. 0 = Fully active, able to carry out all pre-disease activities; 1 = Restricted in strenuous activity but ambulatory and able to carry out work of light or sedentary nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities. Active about 50% of waking hours; 3 = Capable of limited self-care, confined to bed/chair more than 50% of waking hours; 4 = Completely disabled; cannot carry on self-care. Totally confined to bed/chair. 5 = Death.
  Participants
    0 | 1061
    1 | 960
    2 | 197
    3 | 1
    4 | 0
    Missing | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) up to 5 Years
Description: An adverse event (AE) is any untoward medical occurrence in a clinical trial participant regardless of causal relationship to study drug and regardless whether study drug has been administered. A serious adverse event (SAE) is any untoward medical occurrence or effect that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability / incapacity, is a congenital anomaly / birth defect or is medically important due to other reasons than the above mentioned criteria. A non-serious AE is any AE that does not meet the criteria above.
Time Frame: Baseline up to approximately 5 years
Population: Safety set includes all patients who received at least one dose of study drug and had at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | INC424
Number analyzed (Participants) | 2233
Participants
  Adverse Events | 2153
  Serious adverse events | 830

2. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in Spleen Length
Description: Spleen length was assessed by manual palpation. Assessment of spleen response was repeated until early discontinuation of the study drug and also at study completion (28 days post end of treatment visit).
Time Frame: Baseline up to approximately 5 years
Population: Full analysis set includes all patients who received at least one administration of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | INC424
Number analyzed (Participants) | 2049
percentage of participants | 71.7 [69.7 to 73.7]

3. Secondary Outcome: Number of Participants With Best Overall Response (BOR) up to 5 Years According to Spleen Length
Description: Overall response is analyzed using the spleen response, as assessed by the investigator and also by deriving the response using International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria.
  Participants with spleen length at baseline between 5 and 10 cm were reported as Responders if reporting non palpable spleen; Stable disease does not meet criteria for response or disease progression and Progressive disease with an increase of 100% from baseline in spleen length.
  Participants with spleen length at baseline more than 10 cm were reported as Responders with spleen reduction of 50% from baseline; Stable disease does not meet criteria for response or disease progression and Progressive disease with an increase of 50% from baseline in spleen length.
Time Frame: Baseline up to approximately 5 years
Population: Full analysis set includes all patients who received at least one administration of study drug and were observed from baseline in to the study follow-up period.
Measure: Count of Participants; unit: Participants
Groups:
- INC424 - Responders: Responders with spleen length between 5 and 10 cm=non palpable spleen. Responders with spleen length more than 10 cm=Spleen reduction of 50% from baseline.
  5 - 25 mg twice a day (BID) INC424: All patients enrolled into the study will receive INC424 (ruxolitinib). Starting dose is based on baseline platelet counts, with doses ranging from 5 to 20 mg twice a day. No INC424 dose will exceed 25 mg BID orally.
- INC424 - Stable Disease: Participants with Stable Disease with spleen length between 5 and 10 cm=does not meet criteria for response or disease progression.
  Participants with Stable Disease with spleen length more than 10 cm=does not meet criteria for response or disease progression.
  5 - 25 mg twice a day (BID) INC424: All patients enrolled into the study will receive INC424 (ruxolitinib). Starting dose is based on baseline platelet counts, with doses ranging from 5 to 20 mg twice a day. No INC424 dose will exceed 25 mg BID orally.
- INC424 - Progressive Disease: Participants with Progressive Disease with spleen length between 5 and 10 cm=increase of 100% from baseline in spleen length.
  Participants with Progressive Disease with spleen length more than 10 cm=increase of 50% from baseline in spleen length.
  5 - 25 mg twice a day (BID) INC424: All patients enrolled into the study will receive INC424 (ruxolitinib). Starting dose is based on baseline platelet counts, with doses ranging from 5 to 20 mg twice a day. No INC424 dose will exceed 25 mg BID orally.
- INC424 - Missing: Missing values.
  5 - 25 mg twice a day (BID) INC424: All patients enrolled into the study will receive INC424 (ruxolitinib). Starting dose is based on baseline platelet counts, with doses ranging from 5 to 20 mg twice a day. No INC424 dose will exceed 25 mg BID orally.
Arm/Group | INC424 - Responders | INC424 - Stable Disease | INC424 - Progressive Disease | INC424 - Missing
Number analyzed (Participants) | 2178 | 2178 | 2178 | 2178
Participants
  Spleen length at baseline-Less than 5 cm: number analyzed (Participants) | 189 | 189 | 189 | 189
  Spleen length at baseline-Less than 5 cm | NA — Patients with spleen length less than 5 cm are not evaluable (NE) for response. | NA — Patients with spleen length less than 5 cm are not evaluable (NE) for response. | NA — Patients with spleen length less than 5 cm are not evaluable (NE) for response. | NA — Patients with spleen length less than 5 cm are not evaluable (NE) for response.
  Spleen length at baseline-Between 5 and 10 cm: number analyzed (Participants) | 765 | 765 | 765 | 765
  Spleen length at baseline-Between 5 and 10 cm | 421 | 334 | 1 | 9
  Spleen length at baseline-More than 10 cm: number analyzed (Participants) | 1224 | 1224 | 1224 | 1224
  Spleen length at baseline-More than 10 cm | 742 | 463 | 0 | 19

4. Secondary Outcome: Change in Eastern Cooperative Oncology Group (ECOG) Performance Status From Baseline to Worst Post-baseline ECOG Status up to 5 Years
Description: ECOG Performance Score has 5 grades. 0 = Fully active, able to carry out all pre-disease activities; 1 = Restricted in strenuous activity but ambulatory and able to carry out work of light or sedentary nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities. Active about 50% of waking hours; 3 = Capable of limited self-care, confined to bed/chair more than 50% of waking hours; 4 = Completely disabled; cannot carry on self-care. Totally confined to bed/chair. 5 = Death.
Time Frame: Baseline up to approximately 5 years
Population: Full analysis set includes all patients who received at least one administration of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | INC424
Number analyzed (Participants) | 2233
Participants
  Baseline - Grade 0: number analyzed (Participants) | 1061
  Baseline - Grade 0: Worst value post-baseline: Grade 0 | 598
  Baseline - Grade 0: Worst value post-baseline: Grade 1 | 377
  Baseline - Grade 0: Worst value post-baseline: Grade 2 | 62
  Baseline - Grade 0: Worst value post-baseline: Grade 3 | 12
  Baseline - Grade 0: Worst value post-baseline: Grade 4 | 7
  Baseline - Grade 0: Worst value post-baseline: Grade 5 | 0
  Baseline - Grade 0: Worst value post-baseline: Missing | 5
  Baseline - Grade 1: number analyzed (Participants) | 960
  Baseline - Grade 1: Worst value post-baseline: Grade 0 | 89
  Baseline - Grade 1: Worst value post-baseline: Grade 1 | 629
  Baseline - Grade 1: Worst value post-baseline: Grade 2 | 187
  Baseline - Grade 1: Worst value post-baseline: Grade 3 | 26
  Baseline - Grade 1: Worst value post-baseline: Grade 4 | 12
  Baseline - Grade 1: Worst value post-baseline: Grade 5 | 1
  Baseline - Grade 1: Worst value post-baseline: Missing | 16
  Baseline - Grade 2: number analyzed (Participants) | 197
  Baseline - Grade 2: Worst value post-baseline: Grade 0 | 3
  Baseline - Grade 2: Worst value post-baseline: Grade 1 | 43
  Baseline - Grade 2: Worst value post-baseline: Grade 2 | 111
  Baseline - Grade 2: Worst value post-baseline: Grade 3 | 20
  Baseline - Grade 2: Worst value post-baseline: Grade 4 | 12
  Baseline - Grade 2: Worst value post-baseline: Grade 5 | 1
  Baseline - Grade 2: Worst value post-baseline: Missing | 7
  Baseline - Grade 3: number analyzed (Participants) | 1
  Baseline - Grade 3: Worst value post-baseline: Grade 0 | 0
  Baseline - Grade 3: Worst value post-baseline: Grade 1 | 0
  Baseline - Grade 3: Worst value post-baseline: Grade 2 | 0
  Baseline - Grade 3: Worst value post-baseline: Grade 3 | 1
  Baseline - Grade 3: Worst value post-baseline: Grade 4 | 0
  Baseline - Grade 3: Worst value post-baseline: Grade 5 | 0
  Baseline - Grade 3: Worst value post-baseline: Missing | 0
  Baseline - Grade 4: number analyzed (Participants) | 0
  Baseline - Grade 4: Worst value post-baseline: Grade 0 | 0
  Baseline - Grade 4: Worst value post-baseline: Grade 1 | 0
  Baseline - Grade 4: Worst value post-baseline: Grade 2 | 0
  Baseline - Grade 4: Worst value post-baseline: Grade 3 | 0
  Baseline - Grade 4: Worst value post-baseline: Grade 4 | 0
  Baseline - Grade 4: Worst value post-baseline: Grade 5 | 0
  Baseline - Grade 4: Worst value post-baseline: Missing | 0
  Baseline - Missing: number analyzed (Participants) | 14
  Baseline - Missing: Worst value post-baseline: Grade 0 | 1
  Baseline - Missing: Worst value post-baseline: Grade 1 | 8
  Baseline - Missing: Worst value post-baseline: Grade 2 | 4
  Baseline - Missing: Worst value post-baseline: Grade 3 | 1
  Baseline - Missing: Worst value post-baseline: Grade 4 | 0
  Baseline - Missing: Worst value post-baseline: Grade 5 | 0
  Baseline - Missing: Worst value post-baseline: Missing | 0

5. Secondary Outcome: Change in Functional Assessment of Cancer Therapy (FACT-TOI, FACT-G) and FACT-Lymphoma (FACT-Lym) Total Scores Measured at Baseline and Week 48
Description: The FACT-Lym questionnaire consists of a total of 42 questions divided between five subscales (i.e., physical well-being, social/family well-being, emotional well-being, functional well-being and lymphoma subscale). Each subscale questionnaire rates each question on a 5-point scale from 0 = Not at all to 4 = Very much. These scores were summed to three total sum scores, namely FACT-Lym score, FACT-Lym Trial Outcome Index (TOI), FACT-General (FACT-G) and FACT-Lym total score. Total scores: FACT-Lym=0-60, FACT-TOI=0-116, FACT-G total=0-108, FACT-Lym Total= 0-168. Higher scores are reflective of better HRQoL.
Time Frame: Baseline and Week 48
Population: Full analysis set includes all patients who received at least one administration of study drug.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | INC424
Number analyzed (Participants) | 2233
scores on a scale
  FACT-Lymphoma Baseline: number analyzed (Participants) | 2065
  FACT-Lymphoma Baseline | 42.3 (10.20)
  FACT-Lymphoma Week 48: number analyzed (Participants) | 952
  FACT-Lymphoma Week 48 | 47.9 (8.47)
  FACT-Lymphoma TOI Baseline: number analyzed (Participants) | 2034
  FACT-Lymphoma TOI Baseline | 77.9 (18.99)
  FACT-Lymphoma TOI Week 48: number analyzed (Participants) | 940
  FACT-Lymphoma TOI Week 48 | 86.8 (16.42)
  FACT-Lymphoma total score Baseline: number analyzed (Participants) | 2029
  FACT-Lymphoma total score Baseline | 113.9 (24.01)
  FACT-Lymphoma total score Week 48: number analyzed (Participants) | 937
  FACT-Lymphoma total score Week 48 | 123.3 (22.34)
  FACT-G Baseline: number analyzed (Participants) | 2050
  FACT-G Baseline | 71.6 (15.98)
  FACT-G Week 48: number analyzed (Participants) | 950
  FACT-G Week 48 | 75.5 (15.59)

6. Secondary Outcome: Time to First Improvement in FACT-Lym, FACIT-Fatigue Score and ECOG Performance Status
Description: Improvement was defined by the upper limit of the minimally important difference (MID). Patients with the best possible score at Baseline were excluded from this analysis because their HRQoL cannot be further improved. Responders and non-responders for each endpoint were defined based on change from baseline scores using pre specified cut-off points. Patients with an improved score compared to Baseline, for which the magnitude of the change was at least the cutoff value, were classified as responders; otherwise, as non-responders. The responder cutoff: ECOG cutoff=1, range=0 to 5, FACT-Lym cutoff=5.4, range 0-60, FACIT-Fatigue =5 and range=0-52.The median time to first improvement was estimated using the Kaplan Meier method and time to improvement event was determined based on upper bound of the MID. The time to improvement was calculated from the date of first study drug administration.
Time Frame: Baseline up to approximately 5 years
Population: Full analysis set includes all patients who received at least one administration of study drug.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | INC424
Number analyzed (Participants) | 2233
weeks
  FACT-Lym Total score median time to improvement | 10.9 [5.1 to 11.6]
  FACIT - Fatigue score median time to improvement | 4.6 [4.4 to 4.6]
  ECOG score median time to improvement | 63.1 [61.1 to 65.0]

7. Secondary Outcome: Medical Resource Utilization up to 5 Years
Description: Percentage of patients requiring medical resources (blood transfusions, hospitalization, emergency room visits, general practitioners or specialists consultations, urgent care or splenic irradiation) up to 5 years.
Time Frame: Baseline up to approximately 5 years.
Population: Full analysis set includes all patients who received at least one administration of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | INC424
Number analyzed (Participants) | 2233
Participants
  Baseline- Dependency: number analyzed (Participants) | 158
  Baseline- Dependency: End of Study - Dependency | 129
  Baseline- Dependency: End of Study - Independency | 29
  Baseline- Independency: number analyzed (Participants) | 2075
  Baseline- Independency: End of Study - Dependency | 480
  Baseline- Independency: End of Study - Independency | 1595

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected up to 24-months after last patient first visit (LPFV), approximately 5 years .
Description: Safety set includes all patients who received at least one dose of study drug and had at least one post-baseline safety assessment.
  Adverse events occurring more than 28 days after the discontinuation of study treatment are not summarized.
Groups:
- INC424: All patients enrolled into the study will receive INC424 (ruxolitinib). Starting dose is based on baseline platelet counts, with doses ranging from 5 to 25 mg twice a day. No INC424 dose will exceed 20 mg BID orally.
Arm/Group | INC424
All-Cause Mortality (participants affected / at risk) | 205/2233
Serious Adverse Events (participants affected / at risk) | 830/2233
Other Adverse Events (participants affected / at risk) | 2008/2233
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INC424 (N=2233)
Agranulocytosis (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 94
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Bone marrow oedema (Blood and lymphatic system disorders) | 1
Coagulopathy (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Haemolytic anaemia (Blood and lymphatic system disorders) | 2
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1
Hypercoagulation (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 8
Leukostasis syndrome (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Lymphocytosis (Blood and lymphatic system disorders) | 1
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 10
Pancytopenia (Blood and lymphatic system disorders) | 3
Polycythaemia (Blood and lymphatic system disorders) | 1
Splenic haematoma (Blood and lymphatic system disorders) | 3
Splenic infarction (Blood and lymphatic system disorders) | 4
Splenomegaly (Blood and lymphatic system disorders) | 8
Spontaneous haematoma (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 24
Thrombocytosis (Blood and lymphatic system disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 9
Angina pectoris (Cardiac disorders) | 8
Aortic valve incompetence (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 21
Atrioventricular block (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 4
Cardiac arrest (Cardiac disorders) | 16
Cardiac disorder (Cardiac disorders) | 3
Cardiac failure (Cardiac disorders) | 43
Cardiac failure acute (Cardiac disorders) | 5
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 7
Cardiac tamponade (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 9
Cardiogenic shock (Cardiac disorders) | 5
Cardiopulmonary failure (Cardiac disorders) | 1
Conduction disorder (Cardiac disorders) | 1
Congestive cardiomyopathy (Cardiac disorders) | 1
Cor pulmonale (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 5
Coronary artery stenosis (Cardiac disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Intracardiac thrombus (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Left ventricular hypertrophy (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 5
Myocardial ischaemia (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 3
Pericardial haemorrhage (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Right ventricular dysfunction (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 2
Sinus node dysfunction (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 3
Tachyarrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Tricuspid valve incompetence (Cardiac disorders) | 1
Ventricular dysfunction (Cardiac disorders) | 1
Ventricular hypokinesia (Cardiac disorders) | 1
Hydrocele (Congenital, familial and genetic disorders) | 2
Hypoacusis (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 5
Adrenal insufficiency (Endocrine disorders) | 1
Cataract (Eye disorders) | 3
Corneal oedema (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Macular degeneration (Eye disorders) | 1
Optic ischaemic neuropathy (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal mass (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 28
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 5
Abdominal tenderness (Gastrointestinal disorders) | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 2
Anal prolapse (Gastrointestinal disorders) | 1
Anal ulcer (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 14
Barrett's oesophagus (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 17
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Enterovesical fistula (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Femoral hernia (Gastrointestinal disorders) | 1
Gastric haemorrhage (Gastrointestinal disorders) | 4
Gastric stenosis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 21
Haematemesis (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 3
Inguinal hernia (Gastrointestinal disorders) | 5
Inguinal hernia strangulated (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 2
Intestinal infarction (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 4
Mesenteric haemorrhage (Gastrointestinal disorders) | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 2
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Oesophageal haemorrhage (Gastrointestinal disorders) | 2
Oesophageal rupture (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 10
Pancreatitis (Gastrointestinal disorders) | 2
Peritoneal haemorrhage (Gastrointestinal disorders) | 2
Pneumoperitoneum (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3
Rectal polyp (Gastrointestinal disorders) | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 2
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Small intestinal stenosis (Gastrointestinal disorders) | 1
Splenic artery aneurysm (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 3
Tooth loss (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5
Varices oesophageal (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 14
Chest pain (General disorders) | 8
Death (General disorders) | 12
Disease progression (General disorders) | 4
Drug withdrawal syndrome (General disorders) | 2
Face oedema (General disorders) | 1
Fatigue (General disorders) | 11
Gait disturbance (General disorders) | 1
General physical health deterioration (General disorders) | 19
Generalised oedema (General disorders) | 5
Hernia (General disorders) | 1
Hyperpyrexia (General disorders) | 2
Malaise (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 11
Nodule (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 10
Pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Polyp (General disorders) | 1
Pseudocyst (General disorders) | 1
Pyrexia (General disorders) | 79
Sudden death (General disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 2
Biliary colic (Hepatobiliary disorders) | 1
Cholangitis chronic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 3
Cholecystitis acute (Hepatobiliary disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 5
Hepatic failure (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Portal hypertension (Hepatobiliary disorders) | 3
Portal vein thrombosis (Hepatobiliary disorders) | 5
Cytokine release syndrome (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Immunosuppression (Immune system disorders) | 1
Actinomycosis (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 5
Arthritis bacterial (Infections and infestations) | 2
Aspergillus infection (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bacterial infection (Infections and infestations) | 2
Biliary sepsis (Infections and infestations) | 1
Bone tuberculosis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 9
Bronchitis bacterial (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 2
Campylobacter infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 8
Cerebral toxoplasmosis (Infections and infestations) | 1
Community acquired infection (Infections and infestations) | 1
Corneal abscess (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Dermo-hypodermitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Device related sepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 2
Endocarditis (Infections and infestations) | 2
Enterococcal infection (Infections and infestations) | 1
Enterococcal sepsis (Infections and infestations) | 1
Epididymitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 3
Escherichia infection (Infections and infestations) | 2
Escherichia sepsis (Infections and infestations) | 6
Escherichia urinary tract infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 11
Gastroenteritis norovirus (Infections and infestations) | 1
Gastroenteritis salmonella (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 2
Gastrointestinal infection (Infections and infestations) | 3
Genital herpes (Infections and infestations) | 1
H1N1 influenza (Infections and infestations) | 1
Hepatic echinococciasis (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Hepatitis E (Infections and infestations) | 1
Hepatitis infectious (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes simplex pneumonia (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 5
Herpes zoster infection neurological (Infections and infestations) | 1
Infection (Infections and infestations) | 3
Infectious pleural effusion (Infections and infestations) | 1
Influenza (Infections and infestations) | 5
Klebsiella infection (Infections and infestations) | 2
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 3
Lung abscess (Infections and infestations) | 1
Lung infection (Infections and infestations) | 11
Lymph node tuberculosis (Infections and infestations) | 3
Meningitis (Infections and infestations) | 1
Mycobacterial infection (Infections and infestations) | 1
Neurocryptococcosis (Infections and infestations) | 1
Ophthalmic herpes zoster (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 2
Pelvic inflammatory disease (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Peritoneal tuberculosis (Infections and infestations) | 2
Peritonitis (Infections and infestations) | 4
Peritonitis bacterial (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Pneumococcal infection (Infections and infestations) | 1
Pneumocystis jirovecii infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 123
Pneumonia bacterial (Infections and infestations) | 2
Pneumonia pneumococcal (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Pulmonary sepsis (Infections and infestations) | 2
Pulmonary tuberculosis (Infections and infestations) | 2
Pulpitis dental (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Q fever (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 19
Sepsis (Infections and infestations) | 31
Septic shock (Infections and infestations) | 21
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 6
Soft tissue infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 3
Staphylococcal sepsis (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 5
Tubo-ovarian abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 23
Urinary tract infection bacterial (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 8
Vestibular neuronitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Anastomotic leak (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2
Arterial injury (Injury, poisoning and procedural complications) | 1
Brain contusion (Injury, poisoning and procedural complications) | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1
Crush injury (Injury, poisoning and procedural complications) | 1
Face injury (Injury, poisoning and procedural complications) | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 6
Foot fracture (Injury, poisoning and procedural complications) | 2
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 4
Heart injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2
Joint injury (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2
Meniscus injury (Injury, poisoning and procedural complications) | 2
Overdose (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4
Rib fracture (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2
Splenic injury (Injury, poisoning and procedural complications) | 1
Splenic rupture (Injury, poisoning and procedural complications) | 7
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Blast cell count increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 2
Body temperature increased (Investigations) | 1
C-reactive protein increased (Investigations) | 2
Cardioactive drug level increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
Electrocardiogram T wave amplitude increased (Investigations) | 1
Epstein-Barr virus antigen positive (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
General physical condition abnormal (Investigations) | 4
Haemoglobin decreased (Investigations) | 2
Heart rate irregular (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Lipase increased (Investigations) | 1
Myeloblast count increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Portal vein pressure increased (Investigations) | 1
Sensory level abnormal (Investigations) | 1
Transaminases increased (Investigations) | 1
Troponin I increased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 8
Hyperlactacidaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 3
Tumour lysis syndrome (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 11
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic myeloid leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Myeloid metaplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Squamous cell carcinoma of the vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basilar artery aneurysm (Nervous system disorders) | 1
Central nervous system haemorrhage (Nervous system disorders) | 1
Central nervous system lesion (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 4
Coma (Nervous system disorders) | 1
Cranial nerve paralysis (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Drop attacks (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Embolic stroke (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Haemorrhagic stroke (Nervous system disorders) | 2
Headache (Nervous system disorders) | 3
Hepatic encephalopathy (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Hyperaesthesia (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Muscle contractions involuntary (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Neurological decompensation (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 3
Osmotic demyelination syndrome (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Parkinson's disease (Nervous system disorders) | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 11
Transient ischaemic attack (Nervous system disorders) | 5
Device leakage (Product Issues) | 1
Anxiety (Psychiatric disorders) | 1
Anxiety disorder (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 3
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 19
Acute prerenal failure (Renal and urinary disorders) | 1
Anuria (Renal and urinary disorders) | 1
Calculus bladder (Renal and urinary disorders) | 2
Chronic kidney disease (Renal and urinary disorders) | 6
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 6
Nephropathy (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 3
Renal failure (Renal and urinary disorders) | 12
Renal impairment (Renal and urinary disorders) | 2
Renal infarct (Renal and urinary disorders) | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 2
Testicular pain (Reproductive system and breast disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 7
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 36
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 18
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 26
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Panniculitis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Stem cell transplant (Surgical and medical procedures) | 1
Aortic aneurysm (Vascular disorders) | 2
Aortic rupture (Vascular disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Arterial disorder (Vascular disorders) | 2
Arterial haemorrhage (Vascular disorders) | 1
Circulatory collapse (Vascular disorders) | 2
Deep vein thrombosis (Vascular disorders) | 10
Embolism (Vascular disorders) | 1
Haematoma (Vascular disorders) | 9
Hyperaemia (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3
Hypertensive crisis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 7
Pallor (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
Peripheral artery stenosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 3
Phlebitis (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INC424 (N=2233)
Anaemia (Blood and lymphatic system disorders) | 1300
Neutropenia (Blood and lymphatic system disorders) | 146
Thrombocytopenia (Blood and lymphatic system disorders) | 990
Abdominal pain (Gastrointestinal disorders) | 149
Constipation (Gastrointestinal disorders) | 121
Diarrhoea (Gastrointestinal disorders) | 267
Nausea (Gastrointestinal disorders) | 128
Asthenia (General disorders) | 331
Fatigue (General disorders) | 215
Oedema peripheral (General disorders) | 182
Pyrexia (General disorders) | 310
Herpes zoster (Infections and infestations) | 112
Nasopharyngitis (Infections and infestations) | 115
Urinary tract infection (Infections and infestations) | 114
Alanine aminotransferase increased (Investigations) | 134
Platelet count decreased (Investigations) | 198
Weight increased (Investigations) | 140
Arthralgia (Musculoskeletal and connective tissue disorders) | 176
Back pain (Musculoskeletal and connective tissue disorders) | 115
Pain in extremity (Musculoskeletal and connective tissue disorders) | 147
Headache (Nervous system disorders) | 191
Cough (Respiratory, thoracic and mediastinal disorders) | 186
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 155
Pruritus (Skin and subcutaneous tissue disorders) | 131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/14/NCT01493414/SAP_000.pdf
  • Study Protocol (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/14/NCT01493414/Prot_001.pdf